CLINICAL TRIAL: NCT05669859
Title: Efficacy of Postoperative Telerehabilitation in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: karanki1
Record Dates: First submitted 2022-09-12; First posted 2023-01-03 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: adolescent idiopathic scoliosis; telerehabilitation; scoliosis surgery
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The exercise intervention planned in the study includes physical movements and is carried out by connecting to the participant via remote online communication tools.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): It consists of postoperative patients included in the rehabilitation program consisting of approximately one hour of exercise training to be conducted via remote online video-conference (WhatApp Messenger app) for eight weeks, with 2 sessions per week.
  Interventions: Procedure: Exercise
- Control Group (No Intervention): It consists of patients who are called for control by the physician periodically for radiological evaluation and physical examination in the post-surgical period, and who are not included in any rehabilitation program as in routine post-surgical practice.

INTERVENTIONS:
Procedure: Exercise — The rehabilitation program designed in our study was based on the development of core muscle control and dynamic stabilization of the spine, which is generally required by patients. All exercises were combined with controlled breathing, focusing on the mobility of the extremities and the activity of multiple muscle groups.
  Our program created in this direction will start with face-to-face patient education; For 8 weeks, will be carried out remotely online under the supervision of a physiotherapist.On non-telerehabilitation days, they will be asked to keep an exercise diary, instructed to practice the exercise approach presented in sessions at home daily in 20-minute periods. The exercise diary will be checked during online sessions.
  Arms: Telerehabilitation Group

SUMMARY:
In this study, it is aimed to reveal the effects of Tele-Rehabilitation (TR) program, which is designed for the needs of individuals with Adolescent Idiopathic Scoliosis (AIS) who will undergo scoliosis surgery and will be carried out remotely, on pain, trunk endurance, spine flexibility, functional capacity, body appearance perception and quality of life. is intended. With this study, it is aimed to bring evidence-based data on the content of the online rehabilitation program, which can be remotely supervised in the post-surgical period, and the effectiveness and applicability of the applications to the literature.

The study was carried out by Emsey Hospital - Advanced Spine Surgery Unit and Prof. Dr. It is planned with at least 34 individuals with AIS who were treated with Posterior Fusion and Instrumentation technique by an orthopedic specialist at Süleyman Yalçın City Hospital. In the randomized controlled design, experimental type planned study, individuals with a minimum of six months and a maximum of two years after surgery will be divided into two groups as the telerehabilitation group and the control group. Individuals in the telerehabilitation group will be included in the Telerehabilitation program, which is planned as two sessions a week, one to one and a half hours, for eight weeks, via remote online video conferencing method. The control group will not be included in any post-surgery rehabilitation program as it is routinely.

In the study, pain intensity was determined with the "Numerical Rating Scale", body appearance perception with the "Scoliosis Appearance Questionnaire", quality of life with the "SRS-30 Scoliosis Patient Questionnaire", trunk muscle endurance with "position maintenance tests", flexibility of the spine with "Forward Reaching and Side Bending Tests", exercise capacity will be evaluated with the "Six Minute Walking Test". Evaluation of all cases included in the study was planned at two separate times with 8-week intervals. In the analysis of the data, continuous variables will be given as mean ± standard deviation, qualitative variables as number and percentage (%); statistical tests will be determined according to the distribution of the data, and the significance will be taken as p≤0.05 in all measurements.

DETAILED DESCRIPTION:
Scoliosis is a complex three-dimensional deformity characterized by a lateral deviation of the spine of at least 10 degrees in the coronal plane. "Idiopathic Scoliosis", which is the structural and etiological form of scoliosis that develops due to many causes, is called "Adolescent Idiopathic Scoliosis (AIS)" if it occurs in the period from the onset of puberty to the closure of the growth plates.

Current treatment options for scoliosis; It is known as observation, orthosis and surgical intervention, and the choice of the most appropriate treatment depends on the patient's age, menarche status, location and size of the curvature, and risk of progression.

Although children whose curves have reached 40-50 degrees and have not completed their skeletal maturation are generally considered to be indicated for surgical treatment, factors such as the pattern of the curve, the rate of progression, the presence of additional deformity, and failure to respond to conservative treatment also affect the surgical decision. Among the different procedures applied in the surgical treatment of scoliosis, the most frequently applied and effective results of which are shown in the literature is the "Posterior Fusion and Instrumentation" technique. In this technique, motion is eliminated in the relevant segment by fusion to the spine in order to correct the deformity, obtain a balanced spine and prevent the progression of the curvature.

Loss of flexibility and movement in the spine, balance disorder, trunk muscle endurance and a decrease in functional capacity; consequently, the quality of life may deteriorate. In the post-surgical period, it is recommended to rehabilitate the patient under the supervision of a physiotherapist, to provide pain control, to prevent and improve these problems that may occur in the spine.

In the literature, there are deficiencies and lack of evidence in rehabilitative studies after scoliosis surgery. Laurentowska et al. reported that a 4-week endurance training-based rehabilitation program applied 1 to 3 years after surgery provided a significant increase in exercise capacity and emphasized that rehabilitation of patients with scoliosis should be continued after spinal fusion. Weiss found that an in-hospital rehabilitation program based on pain management reduces chronic pain in patients with chronic pain who have had at least 10 years of surgery. In the literature, no sample randomized controlled clinical study was found in which a rehabilitation program was applied to support the adaptation and recovery of the fused spine after scoliosis surgery.

Telerehabilitation is a part of telehealth methods that refers to health care interactions that make use of telecommunications devices in the delivery of traditional face-to-face medical care and processes. It has a wide spectrum and can be defined as "providing rehabilitation services through information and communication technologies". Today, with the development of technological infrastructures, the understanding of telehealth is becoming widespread. Today, the use of telerebilitation is increasing rapidly due to the complexity and difficulty of reaching traditional rehabilitation infrastructures far from where they live, the reduction of hospitalizations and health expenditures, the need for some treatments to be continued for many years, and the ease of communication and organization.

With telerehabilitation, long-distance communication methods can be easily provided through videoconferencing, e-mail and messaging. The use and acceptance of technology by healthcare professionals can help create better quality, safe, successful telerehabilitation programs as a key factor influencing the success and sustainability of telerehabilitation programs.

In the literature, it is seen that telerehabilitation applications give successful results in different patient profiles in individuals with scoliosis who have or have not undergone surgical treatment.

The child with AIS discharged after surgery, both staying away from the medical team and not being able to reach the field-specific health professionals in the area where he lives, may cause him to be deprived of the treatment he needs after the surgery. It is known that today, especially with the effect of the COVID-19 pandemic process, even children, who may have available facilities, do not go to clinics related to contamination risk anxiety and do not receive treatment, as in other patient groups. For all these reasons, conducting treatment programs that will be supervised remotely in safe and effective ways in the post-surgical period can be an effective way to prevent and improve the occurrence of secondary problems after surgery.

In this thesis, it is planned to conduct a live video-conference program under the supervision of a physiotherapist, which is designed in accordance with the recovery processes, needs and literature of individuals with AIS after surgery. With the planned treatment program, it was aimed to investigate the effects of individuals with AIS on postoperative pain, flexibility, trunk muscle endurance, functional capacity, body appearance perception and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be over 9 years old
* Being diagnosed with Adolescent Idiopathic Scoliosis,
* Having been operated with the Posterior Fusion and Instrumentation technique at least 6 months, at most 2 years ago
* Having a device that can be loaded with Internet technology (desktop, laptop, tablet or smartphone)
* Having skills and knowledge about online video communication

Exclusion Criteria:

* Individuals with AIS who have been operated with Anterior or Combined Antero-Posterior Spinal Fusion and Instrumentation, Thoracoscopic Vertebral Body Stretching techniques
* Previous spinal surgery
* Having advanced neuromuscular, rheumatological, orthopedic disease accompanying scoliosis,
* Presence of congenital deformity (short leg, limb agenesis or hypoplasia)
* Having a serious psychiatric or psychological disorder in a medical history,
* Subjected to a separate rehabilitation program accompanied by a physiotherapist,
* Those who are unable to do the evaluation and intervention methods to be applied in the research or who cannot cooperate.
* Individuals who are not suitable to use technological tools and do not have the necessary cognitive skills

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | At the baseline and within one week of completion of the eight-week study period; Change in pain intensity at 8 weeks
  With the Numeric Rating Scale (NRS), the person is asked to mark or say the number corresponding to the subjectively perceived pain intensity (0 = no pain - 10 = unbearable pain) on the scale, using an equally graded linear scale from 0 to 10.
Biering Sorenson Test | At the baseline and within one week of completion of the eight-week study period; Change in trunk extensor muscle endurance at 8 weeks
  It is a valid test that evaluates trunk extensor muscle endurance. The length of time, in seconds, is recorded, when the patient is in the prone position, with the pelvic region and lower extremity in bed, without support.
Kraus Weber testi | At the baseline and within one week of completion of the eight-week study period; Change in trunk flexor muscle endurance at 8 weeks
  It is a valid test that evaluates trunk flexor muscle endurance. While the patient is on the treatment bed, with the hips and knees flexed to 90 degrees, the soles of the feet are fixed on the bed, the body is brought to 60 degrees of flexion and the time that he can stay in this position is recorded in seconds.
Lateral Bridge test | At the baseline and within one week of completion of the eight-week study period; Change in anterior, posterior and lateral stabilizer general muscle endurance at 8 weeks
  It is a valid test used to evaluate anterior, posterior and lateral stabilizer general muscle endurance of the trunk. When the person is in the side-lying position, he is asked to carry his body on his forearms and toes, and the time he can maintain his position is recorded in seconds. Measurements are tested for both sides, right and left.
Forward reach test | At the baseline and within one week of completion of the eight-week study period; Change in flexibility of the thoracolumbar region in the sagittal plane at 8 weeks
  In order to evaluate the flexibility of the thoracolumbar region in the sagittal plane, the patient is asked to lie in a long sitting position, without bending the knees, as far as the arms and feet can reach. The distance between the patient's third hand phalanx and the tips of the toes is measured with a tape measure and recorded in centimeters.
Side bending test: | At the baseline and within one week of completion of the eight-week study period; Change in flexibility of the spine at 8 weeks
  In this test, which is used to evaluate the flexibility of the spine, the patient is standing with his back against the wall, the feet are shoulder-width apart, the arms are on both sides, and the place where the third phalanx touches on the thigh is marked. Then, the patient is asked to bend as far as possible and the difference between the two marks is recorded in centimeters.

SECONDARY OUTCOMES:
Cobb method | At the baseline and within one week of completion of the eight-week study period; Change in curve magnitude at 6 months.
  The Cobb method is the standard measurement method used in coronal grading of the angle of scoliotic curvature on anterior-posterior radiography. On the graph, the angle between the lines drawn parallel to the upper vertebral edge of the curvature at the upper end and the lower edge of the vertebrae at the lower end gives the cobb angle. In order to prevent differences between measurements, measurements will be made by the same researcher with the same equipment.
The Six Minute Walk Test | At the baseline and within one week of completion of the eight-week study period; Change in functional capacity at 8 weeks
  The Six Minute Walk Test is a valid and reliable test used to determine functional capacity. In this test, subjects are asked to walk at the speed they can tolerate best for six minutes in a 30-meter corridor. The distance traveled during this time will be calculated and recorded in meters (m).
Spinal Appearance Questionnaire (Tr-SAQ), | At the baseline and within one week of completion of the eight-week study period; Change in appearance perceptions at 8 weeks
  This questionnaire, with standard drawing images and questions, is a questionnaire designed and developed to measure patients' perceptions and expectations about the appearance of spinal deformities, providing valid and reliable evidence about the anxiety of patients with AIS about the spinal deformity and the development of the curve. Turkish validation was done by Yapar et al.
Scoliosis Research Society Questionnaire- 30 (SRS-30) | At the baseline and within one week of completion of the eight-week study period; Change in quality of life at 8 weeks
  It is a valid and reliable test used to evaluate the health-related quality of life of individuals with scoliosis. It consists of a total of 30 questions, including 5 sub-headings: pain, function, external appearance, mental health and treatment satisfaction. Each question is evaluated out of 5 points, with 1 bad and 5 very good. Turkish validation was performed by Aksekili et al.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Çetinkaya, MSc, Principal Investigator — Haliç University; Tuğba Kuru Çolak, Phd, Study Director — Marmara University; Mehmet Fatih Korkmaz, Phd, MD, Study Chair — İstanbul Medeniyet University; Mehmet Aydoğan, MD, Study Chair — Emsey Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Emsey Hospital, Istanbul
  - Prof. Dr. Süleyman Yalçın City Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No